CLINICAL TRIAL: NCT02984501
Title: Phase II Study of Induction Chemotherapy Followed by Chemoradiotherapy in Patients With Borderline Resectable and Unresectable Locally Advanced Pancreatic Cancer
Brief Title: Study of Induction Chemotherapy Followed by Radiochemotherapy in Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Michele Fiore, MD, Campus Bio-Medico University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20/13 PAR ComEt CBM
Record Dates: First submitted 2016-11-28; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Pancreatic Cancer
Keywords: radiochemotherapy; neoadjuvant therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiation; Neoadjuvant Therapy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Patients treated with induction chemotherapy with gemcitabine and oxaliplatin; for patients without disease progression as detected through restaging exams, chemotherapy was followed by radiochemotherapy which consisted of conformal radiation therapy and concurrent gemcitabine at the dose of 600 mg/mq weekly.
  Interventions: Radiation: Radiation; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Radiation — Radiotherapy target volumes are established by CT scan and PET-CT scan. Radiotherapy is delivered with a total dose of 54-59 Gy with fractionation of 1.8 Gy daily for 5 days a week. The Planning Target Volume (PTV) is defined by CTV with a safety margin of 1cm in all directions to include organ motion and set-up errors. Organs at risk for radiation-induced side effects are contoured on the dose planning CT and dose volume histograms (DVH) are calculated. All treatments are delivered with a 15-MV linear accelerator (Varian Medical System) with a multifield isocentric technique using a multileaf collimator. A quality-control protocol are applied for all patients with periodical digital portal images to evaluate the precision of the set-up.
  Other Names: Neoadjuvant therapy
Drug: Chemotherapy — The induction phase of the treatment plan is designed to administer gemcitabine 1000 mg/mq and oxaliplatin 100 mg/mq every 14 days for four doses. Chemotherapy concurrent to conformal radiation therapy is gemcitabine at the dose of 600 mg/mq weekly.
  Other Names: Induction therapy

SUMMARY:
There is no a clear consensus regarding the optimal treatment of locally advanced pancreatic disease. There is a potential role for neoadjuvant therapy to treat micrometastatic disease with chemotherapy, as well as for the treatment of local disease with radiotherapy. The investigators evaluated the safety and efficacy of induction chemotherapy with oxaliplatin and gemcitabine followed by a high weekly dose of gemcitabine concurrent to radiation therapy in patients with borderline resectable and unresectable locally advanced pancreatic cancer

DETAILED DESCRIPTION:
Continued optimization in multimodality therapy and an accurate patient selection remain crucial points for the appropriate treatment of patients with pancreatic cancer.

In all patients an accurate pre-treatment staging was performed, including: physical examination, complete blood tests and tumor markers, endoscopic ultrasonography (EUS) with fine needle aspiration biopsy, multilayer CT scan, PET-CT (positron emission computed tomography) with 18F-2-fluoro-2-deoxy-D-glucose (FDG) and laparoscopy with peritoneal washing. Jaundiced patients before or during treatment underwent endoscopic biliary stenting.

Patients with the evidence of metastatic disease were excluded, and thus only a small number of patients was consequently enrolled with this neoadjuvant approach.

The induction phase of the treatment plan was designed to administer gemcitabine 1000 mg/mq and oxaliplatin 100 mg/mq every 14 days for four doses.

In the combined phase of the treatment all patients underwent simulation by using a Siemens 16-CT simulator (Siemens Medical System). Radiotherapy target volumes were established by CT scan and PET-CT scan.

Four weeks after the completion of radiochemotherapy, restaging, consisting of clinical examination, laboratory test, tumor markers, CT scan and PET-CT scan, was performed. Tumor response was defined in accordance with the World Health Organization (WHO) definition through CT scan and PET-CT scan. Surgery was considered in patients whose tumors were technically resectable.

After resection, patients were evaluated every three months by means of a standard surveillance protocol that included history and physical examination, cross-sectional imaging and measurement of serum markers, and the intervals were extended to six months after two years

ELIGIBILITY:
Inclusion Criteria:

* proven cytological or histological diagnosis of pancreatic ductal adenocarcinoma;
* borderline resectable or unresectable pancreatic tumours;
* age between 18 and 75 years;
* no previous radiochemotherapy to abdomen;
* 0-I ECOG (Eastern Cooperative Oncology Group) performance status;
* adequate cardiac, liver and kidney function and a good bone marrow reserve.

Exclusion Criteria:

* resectable and metastatic disease;
* previous or concomitant malignant disease;
* one or more of the following clinical conditions: infection, pregnancy or breast-feeding, liver failure, kidney failure, Pa O2 < 65 mmHg, Pa CO2 > 40 mmHg, mental disability.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | four months
  During treatment, patients are evaluated through a directed history, weekly physical examination and blood exams. The occurrence and nature of any adverse events are recorded in accordance with the National Cancer Institute Common Toxicity Criteria (version 4.0) scale. When multiple treatment-related adverse events of the same type occurred in the same patient, only the most severe ones are reported. Subsequently, the dose of chemotherapy is adjusted according to the number of occurrences of grade 2 or greater events.

SECONDARY OUTCOMES:
Overall Survival | 3 years
Progression-free survival | 3 years
metastases-free survival | 3 years
Incidence of Local-regional Tumor Control | 3 years
  Patients are not considered to have local-regional control unless they achieve at least a partial response of their primary tumor or stable disease by imaging. Patients who do not achieve objective response are considered to have local-regional failure. Local-regional control rates are analyzed using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Lucio Trodella, MD, Study Director — Campus Bio-Medico University

IPD SHARING:
Plan to Share IPD: No